CLINICAL TRIAL: NCT04397653
Title: Phase IV Study for Efficacy and Safety of Evolocumab Added to Ezetimibe (Standard of Care) in High Cardiovascular Risk Haemodialized Statin Intolerant Patients With Hypercholesterolemia
Brief Title: Evolocumab Plus Ezetimibe in High Risk Haemodialized Statin Intolerant Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Casilino ASL RMB (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, Professor, Policlinico Casilino ASL RMB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Evolocumab01
Record Dates: First submitted 2020-05-12; First posted 2020-05-21 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Hypercholesterolemia; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: PCSK9 inhibitor; Evolocumab; End-stage renal disease; Hypercholesterolemia; Low-density lipoprotein
MeSH Terms: conditions — Hypercholesterolemia; Kidney Failure, Chronic | interventions — evolocumab; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab + Ezetimibe (Experimental): Patients in this arm will receive subcutaneous evolocumab 140 mg every two weeks plus ezetimibe 10 mg per os daily for 24 weeks
  Interventions: Drug: Evolocumab; Drug: Ezetimibe
- Placebo + Ezetimibe (Placebo Comparator): Patients in this arm will receive subcutaneous placebo every two weeks plus ezetimibe 10 mg per os daily for 24 weeks
  Interventions: Drug: Placebo; Drug: Ezetimibe

INTERVENTIONS:
Drug: Evolocumab — In the intervention arm evolocumab 140 mg subcutaneous every 2 weeks will be administered for 24 weeks to high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia
  Arms: Evolocumab + Ezetimibe
Drug: Placebo — In the placebo arm placebo subcutaneous every 2 weeks will be administered for 24 weeks to high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia
  Arms: Placebo + Ezetimibe
Drug: Ezetimibe — Ezetimibe 10 mg daily will be administered for 24 weeks to high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia in both the placebo arm (plus placebo) and in the intervention arm (plus evolocumab)

SUMMARY:
Evolocumab is a monoclonal antibody that inhibits proprotein convertase subtilisin-kexin type 9 (PCSK9) and lowers low-density lipoprotein (LDL) cholesterol, reducing in turn the risk of cardiovascular events. Whether evolcumab is effective in haemodialized patients is uncertain. The investigators will conduct a randomized, double-blind, placebo-controlled trial to assess the feasibility, safety, and LDL-C-lowering efficacy of evolocumab in high cardiovascular risk haemodialized statin intolerant patients with hypercholesterolemia. Patients will be randomly assigned to receive evolocumab (140 mg subcutaneous every 2 weeks + ezetimibe 10 mg per os daily) or matching placebo (subcutaneous every 2 weeks + ezetimibe 10 mg per os daily) for 24 weeks. The primary efficacy end point will be the reduction in LDL-C ≥ 20 mg/dL from baseline. The key secondary efficacy end points will be: the reduction of LDL-C from baseline at 4, 6 and 12 weeks; the reduction of HDL-C, non-HDL cholesterol and triglycerides from baseline at 24 weeks; the number of patients achieving LDL-C <70 mg/dL. Every adverse event (serious and non-serious) correlated to drug infusion will be recorded (safety end-point).

ELIGIBILITY:
Inclusion Criteria (all of them must be present):

* high cardiovascular risk defined as patients with: Documented cardiovascular disease (CVD), clinical or unequivocal on imaging. Documented clinical CVD includes previous acute myocardial infarction, coronary revascularization and other arterial revascularization procedures, stroke and TIA, aortic aneurysm and PAD. Unequivocally documented CVD on imaging includes plaque on coronary angiography or carotid ultrasound; DM with target organ damage or with a major risk factor such as smoking or marked hypercholesterolaemia or marked hypertension.
* History of statin intolerance, demonstrated by both:

trial of ≥2 statins with intolerance of any dose or to increase statin dose above the total maximum doses because of intolerable: Myopathy or myalgia (muscle pain, ache, or weakness without CK elevation), or Myositis (muscle symptoms with increased CK levels), or Rhabdomyolysis (muscle symptoms with marked CK elevation) and Resolution or improvement of symptoms when the statin dose was decreased or discontinued

* patients with LDL-C ≥70 mg/dL
* end-stage renal disease on chronic hemodialysis

Exclusion Criteria:

* LDL-C <70 mg/dL
* NYHA class III-IV heart failure or last known LVEF <30%
* Uncontrolled serious cardiac arrhythmia, deﬁned as recurrent and highly symptomatic VT, AF with rapid ventricular response, or SVT that are not controlled by medications, within 3 months prior to randomization Planned cardiac surgery or revascularization DM, including: Type 1 DMType 2 DM that is poorly controlled (HbA1c>8.5%) or newly diagnosed within 6 months before randomization; Laboratory evidence of DM during screening (fasting serum glucose ≥126 mg/dL [7.0 mmol/L] or HbA1c≥6.5%) without prior DM diagnosis
* Uncontrolled hypertension, deﬁned as sitting SBP >160mmHg or DBP>100 mm Hg
* Use during the 6 months before LDL-C screening of red yeast rice, niacin >200 mg/d, prescription lipid-regulating drugs (eg, ﬁbrates or derivatives) other than statins, ezetimibe, bile-acid sequestrants, stanols, or stanol esters
* Use during the 12 months before LDL-C screening of a CETP inhibitor such as anacetrapib, dalcetrapib, or evacetrapib
* Use during the 3 months before LDL-C screening of systemic cyclosporine, systemic steroids excluding HRT, vitamin A derivatives (excluding vitamin Ain a multivitamin), or retinol derivatives for the treatment of dermatologic conditions
* Laboratory values at screening TSH < LLN or >1.5 × ULN; CK >3 × ULN; AST or ALT >2 × ULN
* Known concurrent illness within 3 months
* Infection
* Major hematologic, renal, metabolic, GI, or endocrine dysfunction in the judgment of the investigator
* DVT or PE
* Pregnancy, breastfeeding, or inadequate birth control in premenopausal female subjects
* Previous treatment with evolocumab or any other anti-PCSK9 therapy
* Inability to provide informed consent or to attend follow-up visits
* Unreliability as a study participant based on judgment of investigator's knowledge of the subject (eg, alcohol or other drug abuse, inability or unwillingness to adhere to the protocol, psychosis)
* Current enrollment in another investigational device or drug study or <30 d since ending another investigational device or drug study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-11-19 (Estimated); Study Completion 2020-12-14 (Estimated)

PRIMARY OUTCOMES:
LDL cholesterol reduction dichotomic | 24 weeks
  change in LDL cholesterol levels ≥ 20 mg/dL from baseline

SECONDARY OUTCOMES:
LDL cholesterol reduction time-points | 4 weeks, 12 weeks, 24 weeks
  change in LDL cholesterol levels from baseline
HDL cholesterol reduction | 24 weeks
  change in HDL cholesterol levels from baseline
non-HDL cholesterol reduction | 24 weeks
  change in non-HDL cholesterol levels from baseline
Triglycerides reduction | 24 weeks
  change in triglycerides levels from baseline
LDL cholesterol target achieving | 24 weeks
  percent of patients achieving an LDL cholesterol less than 70 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Casilino, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stroes E, Colquhoun D, Sullivan D, Civeira F, Rosenson RS, Watts GF, Bruckert E, Cho L, Dent R, Knusel B, Xue A, Scott R, Wasserman SM, Rocco M; GAUSS-2 Investigators. Anti-PCSK9 antibody effectively lowers cholesterol in patients with statin intolerance: the GAUSS-2 randomized, placebo-controlled phase 3 clinical trial of evolocumab. J Am Coll Cardiol. 2014 Jun 17;63(23):2541-2548. doi: 10.1016/j.jacc.2014.03.019. Epub 2014 Mar 30. PMID 24694531
- [Background] Anderson TJ, Gregoire J, Pearson GJ, Barry AR, Couture P, Dawes M, Francis GA, Genest J Jr, Grover S, Gupta M, Hegele RA, Lau DC, Leiter LA, Lonn E, Mancini GB, McPherson R, Ngui D, Poirier P, Sievenpiper JL, Stone JA, Thanassoulis G, Ward R. 2016 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in the Adult. Can J Cardiol. 2016 Nov;32(11):1263-1282. doi: 10.1016/j.cjca.2016.07.510. Epub 2016 Jul 25. PMID 27712954
- [Background] Expert Dyslipidemia Panel; Grundy SM. An International Atherosclerosis Society Position Paper: global recommendations for the management of dyslipidemia. J Clin Lipidol. 2013 Nov-Dec;7(6):561-5. doi: 10.1016/j.jacl.2013.10.001. Epub 2013 Oct 22. PMID 24314355
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213